CLINICAL TRIAL: NCT00103948
Title: An 18-Week, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Of The Efficacy, Safety, And Tolerability Of Donepezil HCl (E2020) In Patients With CADASIL Who Have Cognitive Impairment
Brief Title: The Efficacy, Safety, And Tolerability Of Donepezil HCl (E2020) In Patients With CADASIL Who Have Cognitive Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2020-A001-233; 2004-001162-40 (EudraCT Number)
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Donepezil

INTERVENTIONS:
Drug: Aricept

SUMMARY:
This is an 18-week, prospective, multi-center, randomized, double-blind, placebo-controlled, (1:1) parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

* Age range - Adult patients, 25 to 70 years of age inclusive
* Gender distribution - Men and women. -- Women of childbearing potential (<1 year postmenopausal) must be practicing effective contraception and have a negative serum bHCG at Screening. Pregnant and/or lactating females are excluded. Patients who become pregnant during the study will be discontinued.
* Diagnostic evidence of CADASIL either by (1) identification of a NOTCH3 mutation (excluding polymorphisms) or (2) presence of typical deposits on an electron microscopy of a skin biopsy.
* Cognitive impairment - (1) Subjects or their study partners must give a description of cognitive problems and one of the following: (2a) MMSE score of 10-27 (inclusive) or (2b) Trails B score, 1.5 standard deviations below the mean after adjustment for age and education.
* Head MRI - Evidence of disease consistent with CADASIL, and no evidence of another disease, which might account for cognitive impairment or dementia (as judged by the Investigator/physician at the site). (The latter may be determined with a CT head scan for eligibility purposes. The MRI would still be needed.) Must be obtained within 6 months of the Screening/Baseline visit. If no such head MRI had been previously obtained, a head MRI will be obtained as part of Screening/Baseline after all other inclusion and exclusion criteria (except clinical laboratory determinations) are satisfied. Patients in whom an MRI is contraindicated can have a CT instead, however, MRI is the preferred modality.
* Race and ethnicity - Any race and ethnic group.
* Health - Generally healthy, ambulatory or ambulatory-aided (i.e., walker, cane or wheelchair) outpatient. Speech, motor function, comprehension, and corrected vision and hearing must be sufficient for compliance with all testing procedures.
* Clinical laboratory values must be within normal limits, or if abnormal, must be judged clinically insignificant by the Investigator/ physician.
* Patients with Vitamin B12 deficiency who are on a stable dose of medication for at least 12 weeks prior to Screening/Baseline and who have normal serum B12 levels at Screening/ Baseline will be eligible. Patients who might otherwise have been eligible can be re- screened when they meet this criterion. This stable dose of Vitamin B12 must be maintained throughout the study.
* Patients with hypothyroidism or hyperthyroidism who are on a stable dose of medication for at least 12 weeks prior to Screening, have a normal TSH and free T4 at screening, and are considered euthyroid will be eligible. Patients who might otherwise have been eligible can be re-screened when they meet this criterion. This stable dose must be maintained throughout the study.
* Patients must have a reliable study partner who has regular contact with the patient (e.g., an average of 4 or more contacts per week), can observe for possible adverse events, and can accompany the patient to all visits.
* Patients with a history of hypertension, cardiac disease, diabetes, or peripheral vascular disease, may be enrolled in the study provided that the following standards are met. -- Hypertension must be medication controlled (sitting SBP < 175, sitting DBP < 100 mm Hg) and cardiac disease (e.g., angina pectoris, congestive heart failure, right bundle branch block, or arrhythmias) is stable on appropriate medication for 12 weeks prior to Screening.

Peripheral vascular disease must have been stable for 12 weeks prior to Screening. No elective surgical procedures should be planned during the course of the study (e.g., hernia repair and bunion removal). Patient with diabetes must be stable as demonstrated by an HbA1c of <= 8.0% or a random serum glucose value of <= 170 mg/dL.

* All patients with CADASIL are at risk for stroke/TIA and may be enrolled in the study provided that no new strokes have been diagnosed or identified to have occurred within the three months prior to Screening. Patients who might otherwise be eligible can be screened 12 weeks after the stroke. Patients with TIAs are eligible without a waiting period. Patients who are already enrolled will continue in the study as assessed by the Investigator/ physician.
* Patients with CADASIL may suffer depression. Such patients are eligible for enrollment if they are stable on medication for 12 weeks and have an MADRS score < 20. Patients with an MADRS score >= 20 may be re-screened after 12 weeks on a stable dose of medication. This stable dose must be maintained throughout the study.
* Minor medical conditions must be stable before study enrollment.
* Patients who are taking Gingko Biloba or Vitamin E and have been taking stable doses of these compounds for 8 weeks are allowed in the study. This stable dose must be maintained throughout the study.

Exclusion Criteria:

* Neurological disorders affecting cognition or the ability to assess it that are not associated with CADASIL, such as Alzheimer's Disease, Parkinson's disease, normal pressure hydrocephalus, idiopathic seizure disorders, multiple sclerosis, cerebral vasculitis or infections of the central nervous system, subdural hematoma, as well as Human Immunodeficiency Virus (HIV) disease, a history of significant head trauma followed by persistent neurological deficits, sleep disorders affecting level of consciousness, or known structural brain abnormalities.
* Psychiatric disorders affecting the ability to assess cognition that are not typically associated with CADASIL, such as schizophrenia.
* Active drug or alcohol abuse or dependence in <= 5 years by DSM-IV criteria.
* Any active or clinically significant conditions affecting absorption, distribution, or metabolism of the study medication (e.g., inflammatory bowel disease, hepatic disease, or severe lactose intolerance).
* Uncontrolled hypertension (sitting systolic >= 175 mmHg and/or diastolic >= 100 mmHg) as assessed by the Investigator regardless of whether the patient is taking antihypertensive medication.
* Evidence of clinically significant, active gastrointestinal, renal, hepatic, respiratory, infectious, endocrine, or cardiovascular system disease. A patient so excluded, who subsequently becomes stable for 4 weeks, may become eligible for enrollment if Inclusion Criteria 2) and 3) are met.
* Patients with left bundle branch block are excluded.
* History of malignant neoplasms (does not include basal or squamous cell carcinoma of the skin) treated within 2 years prior to study entry, current evidence of malignant neoplasm, or recurrent or metastatic disease.
* Women who are pregnant or breastfeeding.
* Patients and/or study partners who are unwilling or unable to fulfill the requirements of the study.
* Known hypersensitivity to cholinesterase inhibitors or piperidine-containing drug.
* Use of any unapproved prior or concomitant medications as defined in the protocol.
* Any condition that would make the patient or study partner, in the opinion of the Investigator, unsuitable for the study.
* Involvement in any other investigational trial in the preceding 12 weeks or likely involvement in any other investigational study drug trial during the course of this study. Prior to enrollment, the study director or medical monitor must approve involvement in investigational trials that do not involve a study drug.
* Patients with changes in doses of concomitant medication, not otherwise described, within the 6 weeks prior to enrollment.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2005-02; Primary Completion 2006-10 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Moline, Ph.D., Study Director — Eisai Inc.
Locations (4):
- United States (2):
  - Jose Biller, M.D., Maywood, Illinois
  - New York University School of Medicine, New York, New York
- Woodville, South Australia, Australia
- Málaga, Spain

REFERENCES:
- [Derived] Dichgans M, Markus HS, Salloway S, Verkkoniemi A, Moline M, Wang Q, Posner H, Chabriat HS. Donepezil in patients with subcortical vascular cognitive impairment: a randomised double-blind trial in CADASIL. Lancet Neurol. 2008 Apr;7(4):310-8. doi: 10.1016/S1474-4422(08)70046-2. Epub 2008 Feb 28. PMID 18296124